CLINICAL TRIAL: NCT06519851
Title: Combined Shoulder Anterior Capsule and Suprascapular Nerve Block Versus Interscalene Block in Shoulder Surgery: Randomized Controlled Clinical Trial
Brief Title: Combined Shoulder Anterior Capsule and Suprascapular Nerve Block Versus Interscalene Block in Shoulder Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Abbas, assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHAC & SSNB
Record Dates: First submitted 2024-07-06; First posted 2024-07-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Bupivacaine; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • SSNB & SHAC (Active Comparator): patients will receive general anesthesia + ultrasound guided suprascapular nerve block (SSNB) with 10 ml bupivacaine 0.25% deep to the transverse scapular ligament and Shoulder anterior capsule (SHAC) block with 30 ml bupivacaine 0.25% (20 ml deep to the deltoid muscle between the deltoid and subscapularis tendon &10mL in the pericapsular space)
  Interventions: Other: suprascapular nerve block with 10 ml bupivacaine 0.25% & shoulder anterior capsule block with 30 ml bupivacaine 0.25%
- • Interscalene (Placebo Comparator): patients will receive general anesthesia + ultrasound guided interscalene brachial plexus block (ISB) with 20 ml bupivacaine 0.25% around C5-C6-C7 nerve roots of the brachial plexus.
  Interventions: Other: Interscalene block with 20 ml bupivacaine 0.25%

INTERVENTIONS:
Other: suprascapular nerve block with 10 ml bupivacaine 0.25% & shoulder anterior capsule block with 30 ml bupivacaine 0.25% — postoperative analgesic effect of combined shoulder anterior capsule (SHAC) block with suprascapular nerve block (SSNB) following shoulder surgery by ultrasound guided suprascapular nerve block (SSNB) with 10 ml bupivacaine 0.25% deep to the transverse scapular ligament and Shoulder anterior capsule (SHAC) block with 30 ml bupivacaine 0.25% (20 ml deep to the deltoid muscle between the deltoid and subscapularis tendon &10mL in the pericapsular space)
  Arms: • SSNB & SHAC
Other: Interscalene block with 20 ml bupivacaine 0.25% — postoperative analgesic effect of Interscalene block (ISB) following shoulder surgery by ultrasound guided interscalene brachial plexus block (ISB) with 20 ml bupivacaine 0.25% around C5-C6-C7 nerve roots of the brachial plexus
  Arms: • Interscalene

SUMMARY:
The study aims to evaluate the postoperative analgesic effect of combined shoulder anterior capsule (SHAC) block with suprascapular nerve block (SSNB) versus Interscalene block (ISB) during the first 24 hours following shoulder surgery.

DETAILED DESCRIPTION:
Significant acute postoperative pain is common in adults after shoulder surgery, with approximately 45% reporting severe pain in the immediate postoperative period. This pain may necessitate opioid use for several days. The opioid requirement may be similar to that following gastrectomy or thoracotomy, and opioid-only analgesic techniques for shoulder surgery are commonly associated with opioid-related adverse effects such as nausea , vomiting, respiratory depression, pruritus, allergic reactions, sleep disturbance and constipation.

With the majority of these procedures being performed in the ambulatory setting, providing effective postoperative analgesia has become paramount in promoting quicker recovery and rehabilitation of these patients. Thus, alternative techniques are preferred. Nowadays, several ultrasound guided regional anesthesia methods are used for postoperative analgesia .

The shoulder is formed by two joints the acromioclavicular joint formed by the acromion process of the scapula and the clavicle, and the glenohumeral joint formed by the glenoid process of the scapula and the humeral head.

The shoulder joint is innervated by branches of the brachial plexus which include the suprascapular nerve, the axillary nerve, the subscapularis and lateral pectoral nerves .

The suprascapular nerve arises from the ventral rami of cervical nerve roots (C5 and C6), and it is a branch of the superior trunk of the brachial plexus. The suprascapular nerve is a mixed motor and sensory nerve providing motor innervation to the supraspinatus and infraspinatus muscles. And sensory innervation to the acromioclavicular joint, glenohumeral joint, and ligaments of the shoulder. The axillary nerve also originates from the ventral rami of C5 and C6 and it is a terminal branch of the brachial plexus. The axillary nerve is a mixed motor and sensory nerve providing motor innervation to the deltoid and sensory contributions to the glenohumeral joint . Other nerves involved in the sensory innervation of the shoulder joint include the nerve to subscapularis and the lateral pectoral nerve both of which arise from ventral rami of C5 and C6.

Cutaneous innervation is also important to consider in performing regional anesthesia. The cutaneous innervation of the shoulder is provided by branches of the brachial plexus with minor contributions from thoracic nerve roots. The supraclavicular nerve arises from cervical 3 and 4 nerve roots and provides cutaneous innervation to the cape of the shoulder. The axillary nerve provides cutaneous innervation over the lateral aspect of the shoulder.

Interscalene block which anesthetizes C5 and C6 nerve roots is the gold standard regional anesthesia technique for shoulder surgery but it carries a risk of ipsilateral phrenic nerve block and hemidiaphragmatic paralysis which limit its use in patients with preexisting pulmonary compromise. Less common complications included respiratory distress, weakness of the arm, hoarseness of voice, Horner's syndrome and brachial plexus neuropathy, rebound pain, and pneumothorax.Therefore, selecting the most appropriate brachial plexus block method is crucial to achieve effective pain control avoid complications.

Various diaphragm-sparing alternatives to interscalene blocks have been studied. Among them is the suprascapular nerve block (SSNB) which accounts for about 70% of the sensory innervation of the shoulder. Consequentially, it has been suggested that the SSNB will deliver adequate analgesia for shoulder surgery, but sometimes does not provide adequate analgesia because the axillary nerve, the lateral pectoral nerve, and sometimes the musculocutaneous nerve also contribute to the complex innervation of the shoulder joint.

By combining the (SSNB) with a recently described new block, the shoulder anterior capsular block (SHAC) , the investigator can reach all our targets. The SHAC is the combination of two different blocks. The first block is via the interfacial space between the deep layer of the deltoid fascia and the superficial layer of the subscapularis fascia, anterior to the subscapularis myotendinous junction, we can block both the axillary nerve and the subscapular nerves, the lateral pectoral nerve, and the musculocutaneous nerve. Second block, Pericapsular nerve group block (PENG) which is based in permeable spaces between the three glenohumeral ligaments as potential gateways. For example, it was suggested that deep pericapsular infiltration of local anesthetic towards the subscapularis may cover the axillary and subscapularis branches that feed the anteroinferior and superior quadrants of the glenohumeral joint by injecting the pericapsular space, reaching the terminal articular branches indistinctly from their origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* patients aged 18-65 years
* BMI of less than 30
* American Society of Anesthesiologists (ASA) physical status I-II,
* Patients scheduled for unilateral shoulder surgery under general anesthesia.

Exclusion Criteria:

* Patient refusal
* BMI of 30 or more
* ASA III or more
* Pregnancy or breast feeding
* Uncooperative patients with communication difficulties, which might prevent a reliable postoperative assessment.
* Shoulder revision surgery
* Pre-existing neurological deficits or neuropathy
* Known contraindications to peripheral nerve block, including local skin infections in the block procedure area, bleeding diathesis, coagulopathy
* Patients with chest problems not eligible for ISB

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative analgesia measured by Visual analogue scale during the first 24 hours after shoulder surgery. | Pain will be assessed at 1st hour, then at 2, 6, 12, 18 and 24 hours postoperatively using VAS score.
  Visual analogue scale consists of a 10 centimeter line, with two end points representing 0 (no pain) and 10 (worst imaginable pain)

SECONDARY OUTCOMES:
The first time to rescue opioid analgesia, and the total opioid consumption in the first 24 hours postoperatively | 24 hours postoperatively
  The first time to rescue opioid analgesia, and the total opioid consumption in the first 24 hours postoperatively
Any Complications related to the blocks | 24 hours postoperatively
  Any Complications related to the blocks as hemodynamic changes, hoarseness of voice, Horner syndrome, vascular injury, sensory or motor side effects.